CLINICAL TRIAL: NCT04593628
Title: Adapting 'Connect for Caregivers' for Hispanic Caregivers: A Pilot Study for Year Two of the Rochester Roybal Center for Social Ties and Aging Research (P30AG064103) and the UR Healthy Aging Research Program (HARP)
Brief Title: Connection for Latinos Caring for a Loved One With Dementia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study aims changed based on the results of a earlier qualitative study.
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Caroline Silva, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005437; P30AG064103 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Social Isolation; Loneliness
MeSH Terms: conditions — Social Isolation | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental)
  Interventions: Behavioral: Connect for Caregivers

INTERVENTIONS:
Behavioral: Connect for Caregivers — The STAR Center developed Connect for Caregivers to help improve connectedness among older caregivers of individuals with Alzheimer's Disease and Related Dementias (ADRD). Connect for Caregivers includes three components: (1) psychoeducational materials on the importance of connectedness for health and well-being; (2) a card sort-based 'discussion prioritization tool' that systematizes and routinizes the process of identifying and prioritizing barriers to connectedness; (3) personalized resources to address the identified barriers/targets. We will tailor Connect for Caregivers for Hispanic/Latino and Spanish-speaking caregivers guided by the Selective and Directed Treatment Adaptation Framework. The intervention is given once during the study.

SUMMARY:
The purpose of this research study is to culturally adapt a personalized intervention for Hispanic/Latino caring for a loved one with significant memory problems. The intervention will be designed to help Hispanics/Latinos caring for a loved one with significant memory problems in their own unique context to: 1.) understand the importance of social connections for their own health and well-being, 2.) learn to become aware of their own personal barriers to social connections, and 3.) increase their knowledge of local resources for promoting social connections.

ELIGIBILITY:
Inclusion Criteria:

* Current or previous Hispanic/Latino caregiver (English or Spanish speaking) for a community-dwelling loved one with ADRD, living with (or in close proximity to) loved one with dementia;
* Age 40 or older;
* Able to provide informed consent to participate in the research study.

Exclusion Criteria:

* Primary language is not English or Spanish;
* Current alcohol or substance abuse, psychotic disorders (current and lifetime), bipolar disorder and current mood disorders with psychotic features (MINI International Neuropsychiatric Interview);
* Significant cognitive impairment on a cognitive screening measure at the HARP screening assessment (Telephone Interview for Cognitive Status; TICS < 25);
* Hearing problems that preclude completion of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Basic Psychological Need Satisfaction at Post Intervention | Baseline and 1 hour
  The Basic Psychological Need Satisfaction and Frustration Scales (BPNSFS) will be used. The BPNSFS consists of 24 items assessing both satisfaction and frustration in the need for competence, autonomy, and relatedness, as posited by Self-Determination Theory. We will report changes in the three BPNSFS subscales measuring satisfaction in: autonomy, relatedness and competence. Items are scored on a 1-5 Likert scale with each subscale score ranging from 4-20. Higher scores indicating greater satisfaction. Mean change in subscale scores (change = post intervention scores - baseline scores) will be reported.
Change from Baseline in Basic Psychological Need Frustration at Post Intervention | Baseline and 1 hour
  The Basic Psychological Need Satisfaction and Frustration Scales (BPNSFS) will be used. The BPNSFS consists of 24 items assessing both satisfaction and frustration in the need for competence, autonomy, and relatedness, as posited by Self-Determination Theory. We will report changes in the three BPNSFS subscales measuring frustration in: autonomy, relatedness and competence. Items are scored on a 1-5 Likert scale with each subscale score ranging from 4-20. Higher scores indicating greater frustration. Mean change in subscale scores (change = post intervention scores - baseline scores) will be reported.
Change from Baseline in Ability to Participate in Social Roles and Activities at Post Intervention | Baseline and 1 hour
  The PROMIS Ability to Participate in Social Roles and Activities measure will be used. This scale assesses the perceived ability to perform one's usual social roles and activities. The scale is administered as a computerized adaptive test (CAT) based on a 35 item bank; items are scored on a 1-5 Likert scale. Items are worded negatively in terms of perceived limitations, but responses are reverse-coded. CAT raw scores are converted into T-scores (0-100), with higher scores representing fewer limitations (better abilities). Mean change in T-scores (change = post intervention scores - baseline scores) will be reported.

SECONDARY OUTCOMES:
Change from Baseline in General Self-Efficacy Score at Post Intervention | Baseline and 1 hour
  The PROMIS General Self-Efficacy measure will be used. This scale assesses confidence in one's ability to perform specific tasks or behaviors. The scale is administered as a computerized adaptive test (CAT) based on a 10 item bank; items are scored on a 1-5 Likert scale. CAT raw scores are converted into T-scores (0-100), with higher scores indicating greater self-efficacy. Mean change in T-scores (change = post intervention scores - baseline scores) will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No